CLINICAL TRIAL: NCT04139525
Title: Comparison of Citrate and Heparin Anticoagulation During Hemodialysis With Medium Cut-off Polyarylethersulphone- Polyvinylpirrolidone (Theranova) Membrane
Brief Title: Comparison of Citrate and Heparin Anticoagulation During Hemodialysis With MCO PES-PVP (Theranova) Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marija Malgaj Vrečko (Other)
Responsible Party: Sponsor-Investigator, Marija Malgaj Vrečko, Principal Investigator, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0120-11/2019/3
Record Dates: First submitted 2019-10-12; First posted 2019-10-25 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: End Stage Renal Disease; Haemodialysis; Anticoagulation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Heparin; trisodium citrate

STUDY DESIGN:
Intervention Model Description: The research will be performed as a prospective clinical trial. Every patient will have 2 HD procedures with PES-PVP membrane in a randomized order: 1 with unfractionated heparin (UFH) and 1 with 8% trisodium citrate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unfractionated heparin and 8% trisodium citrate (Experimental): Unfractionated heparin and 8% trisodium citrate.
  Interventions: Biological: unfractionated heparin; Biological: 8% trisodium citrate

INTERVENTIONS:
Biological: unfractionated heparin — A bolus of 30 I.U./kg at the start of hemodialysis, followed by 18 I.U./kg per every hour of hemodialysis.
Biological: 8% trisodium citrate — 8% trisodium citrate in the dose of 150 ml/h.

SUMMARY:
The purpose of the study is to compare the efficiency and biocompatibility of citrate and heparin anticoagulation during hemodialysis with medium cut-off polyarylethersulphone-polyvinylpirrolidone membrane (Theranova®).

DETAILED DESCRIPTION:
The purpose of the study is to compare the efficiency and biocompatibility of citrate and heparin anticoagulation during hemodialysis (HD) with PES-PVP membrane. The research will be performed as a prospective clinical trial and will include 35 patients. Every patient will have 2 HD procedures with PES-PVP membrane in a randomized order: 1 with unfractionated heparin (UFH) and 1 with 8% trisodium citrate. We will compare the efficiency of both types of anticoagulation by measuring overall and instantaneous clearances of small, middle and protein-bound molecules (urea, creatinine, phosphate, β2-microglobulin, p-cresol). Biocompatibility will be evaluated by measuring activation of: complement (serum concentration of C3a and C5a), leukocytes (serum concentration of myeloperoxidase) and thrombocytes (serum concentration of PF4). We will also monitor complete blood count for occurrence of leukopenia and thrombocytopenia. After the HD electron microscopy of the membrane will be done in the proportion of included patients to evaluate adsorption of cells and formation of blood clots on the membrane.

ELIGIBILITY:
Inclusion Criteria:

* patient on chronic hemodialysis
* age 18 years old or more
* being able to give an informed consent to participate in the survey

Exclusion Criteria:

* on therapeutic anticoagulation
* citrate or heparin contraindicated
* citrate or heparin intolerance
* acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clearance of beta-2 microglobulin | At the end of each hemodialysis procedure.
  Overall and instantaneous clearance of beta-2 microglobulin.
Clearance of phosphate | At the end of each hemodialysis procedure.
  Overall and instantaneous clearance of phosphate.
Serum concentration of C3a, C5a, myeloperoxidase and PF-4 | At the start, after 15 minutes and at the end of each hemodialysis procedure.
  Blood for the laboratory measurements will be taken from the arterial line.

SECONDARY OUTCOMES:
Clearance of urea | At the end of each hemodialysis procedure.
  Overall and instantaneous clearance of urea.
Clearance of creatinine | At the end of each hemodialysis procedure.
  Overall and instantaneous clearance of creatinine.
Clearance of p-cresol | At the end of each hemodialysis procedure.
  Overall and instantaneous clearance of p-cresol.
White blood cell count | At the start, after 15 minutes and at the end of each hemodialysis procedure.
  Blood for the laboratory measurements will be taken from the arterial line.
Blood platelet count | At the start, after 15 minutes and at the end of each hemodialysis procedure.
  Blood for the laboratory measurements will be taken from the arterial line.

CONTACTS AND LOCATIONS:
Overall Officials: Marija Malgaj Vrečko, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vrecko MM, Pajek J, Buturovic-Ponikvar J. Use of regional citrate anticoagulation with medium cut-off membrane: pilot report. BMC Nephrol. 2022 Oct 27;23(1):346. doi: 10.1186/s12882-022-02960-y. PMID 36303108